CLINICAL TRIAL: NCT06668142
Title: A Prospective, Multicenter, Open-label Study of the Beacon Platform for Holmium Laser Enucleation of the Prostate (HoLEP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andromeda Surgical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTRA112024
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: HoLEP; RoLEP; Robotic HoLEP; BPH; Prostate; urology; robotic; Andromeda; ASTRA
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A single-arm open label pilot study (Experimental): A single-arm open label pilot study observing intraoperative and postoperative outcomes of the Beacon Platform in HoLEP.
  Interventions: Device: Beacon Platform

INTERVENTIONS:
Device: Beacon Platform — The Beacon Platform is a robotically assisted surgical (RAS) device. It enables the urologist, through software, to control and move surgical instruments for a variety of transurethral, endoscopic procedures

SUMMARY:
Robotic assisted surgery for benign prostatic hyperplasia (BPH)

DETAILED DESCRIPTION:
A single-arm open label pilot study observing intraoperative and postoperative outcomes of the Beacon Platform in HoLEP.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Subject has diagnosis of lower urinary tract symptoms and/or urinary retention due to benign prostatic enlargement causing bladder outlet obstruction,
3. Subject is able and willing to comply with all the assessments of the study,
4. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate, and has signed the informed consent form,
5. ≥ 45 years of Age,
6. Prostate volume 40 - 120 cc by transrectal ultrasound (TRUS), magnetic resonance imaging (MRI), or computed tomography (CT), measured within one year prior to procedure,
7. The subject is indicated for undergoing HoLEP procedure

Exclusion Criteria:

1. Urethral stricture, meatal stenosis, or bladder neck contracture - either current or recurrent,
2. History of prostate cancer or current/suspected bladder cancer,
3. Prostate cancer should be ruled out before participation to the satisfaction of the investigator if Prostate-Specific Antigen (PSA) is above acceptable thresholds,
4. History of other diseases causing voiding dysfunction including urinary retention (e.g., diagnosis of neurogenic bladder, Parkinson's disease, multiple sclerosis, etc.),
5. Subjects with overactive bladder in the absence of benign prostatic obstruction as determined by the investigator,
6. Acute urinary tract infection (UTI) or finding of asymptomatic bacteriuria (Note: subject can be enrolled if the UTI is treated)
7. Previous pelvic irradiation or radical pelvic surgery,
8. Previous prostate surgery, including enucleation, resection, vaporization, thermotherapy, ablation, stenting, or prostatic urethral lift,
9. Inability to stop taking anticoagulants for at least 3 days prior to the procedure or antiplatelets and/or coumadin for at least 5 days prior to the procedure (Note: low dose aspirin therapy is permitted),
10. Any severe illness that would prevent complete study participation or confound study results.
11. Bleeding tendency disorders,
12. Future fertility concerns,
13. Subject has any other disease or condition(s) that would interfere with completion of the study and follow-up assessments, would increase risks of the procedure, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect outcomes,
14. Concomitant participation in another interventional study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Any potential participants who were assigned male at birth (ie have a prostate) but do not identify as male may still participate.
Enrollment: 54 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Successfully Completing Robot-Assisted HoLEP (Enucleation and Morcellation) Without Conversion | During the procedure.
  This endpoint measures the number of participants who successfully complete both the enucleation and morcellation phases of robot-assisted HoLEP (Holmium Laser Enucleation of the Prostate) without the need to convert to a conventional HoLEP or an alternative surgical procedure for treating BPH-related LUTS.Successful completion is defined as completing both phases without using additional devices .
  This excludes the Roll-in subjects and the use of other devices for hemostasis or dissecting the enucleated tissue during or after the procedure.
Number of subjects with adverse events ( Clavien-Dindo Grade 3a or higher ) | From procedure date to 30 days
  Proportion of subjects with adverse events rated as probably or definitely related to the study procedure (robot-assisted HoLEP or RoLEP) classified as Clavien-Dindo Grade 3a or higher through 30 days post-treatment.

SECONDARY OUTCOMES:
Number of Participants with Capsular Perforation Leading to Procedure Interruption or Conversion | From procedure date to 30 days.
  This outcome measures the incidence of capsular perforation events that result in interruption of the procedure or conversion to conventional HoLEP or an alternative surgical procedure
Number of Participants with Bladder Perforation Leading to Procedure Interruption or Conversion | From procedure date to 30 days.
  This outcome measures the incidence of bladder perforation events that result in interruption of the procedure or conversion to conventional HoLEP or an alternative surgical procedure.
Number of Participants with Ureteric Orifice Damage Requiring Intervention | From procedure date to 30 days.
  This outcome assesses the incidence of ureteric orifice damage leading to stricture, stenting, or any other sequelae or subsequent intervention.
Length of Hospital Stay Post-Procedure | From procedure date to 30 days
  This outcome measures the total length of hospital stay required following the HoLEP procedure.
Length of Catheterization Post-Procedure | From procedure date to 30 days
  This outcome measures the total duration of catheterization following the procedure.
Operative Time for Procedure Completion | During the procedure.
  This outcome measures the total time required to complete the HoLEP procedure.
Number of Participants with Repeat Hospitalization for Genitourinary Conditions | From procedure date to 30 days post-procedure.
  This outcome measures the incidence of repeat hospitalizations due to genitourinary conditions within 30 days post-procedure.

OTHER OUTCOMES:
Duration of Enucleation and Morcellation Phases | During the procedure.
  This outcome measures the combined time taken to complete the enucleation and morcellation phases of the HoLEP procedure.
Number of Participants Requiring Blood Transfusion Post-Procedure | From procedure date to 30 days.
  This outcome tracks the incidence of blood transfusion events following the HoLEP procedure.
Number of Participants Requiring Secondary Reintervention with HoLEP or Alternative Surgical Therapy | From procedure date to 30 days.
  This outcome measures the incidence of participants requiring a secondary reintervention using HoLEP or an alternative surgical therapy for LUTS within 30 days post-procedure.
Incidence Rate of Stress Urinary Incontinence Post-Procedure | From procedure date to 30 days.
  This outcome assesses the rate of stress urinary incontinence among participants within 30 days following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gilling, MD, FRACS, Principal Investigator — Tauranga urology research; Rodrigo Ledezma, MD,, Principal Investigator — University of Chile Clinical Hospital
Locations (3):
- Chile (2):
  - Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Hospital Clínico de la Universidad de Chile, Santiago, Santiago Metropolitan
- Tauranga Urology Research Limited, Tauranga, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shvero A, Kloniecke E, Capella C, Das AK. HoLEP techniques - lessons learned. Can J Urol. 2021 Aug;28(S2):11-16. PMID 34453423
- [Background] Abedi A, Razzaghi MR, Rahavian A, Hazrati E, Aliakbari F, Vahedisoraki V, Allameh F. Is Holmium Laser Enucleation of the Prostate a Good Surgical Alternative in Benign Prostatic Hyperplasia Management? A Review Article. J Lasers Med Sci. 2020 Spring;11(2):197-203. doi: 10.34172/jlms.2020.33. Epub 2020 Mar 15. PMID 32273963
- [Background] Das AK, Han TM, Hardacker TJ. Holmium laser enucleation of the prostate (HoLEP): size-independent gold standard for surgical management of benign prostatic hyperplasia. Can J Urol. 2020 Aug;27(S3):44-50. PMID 32876002
- [Background] Das AK, Teplitsky S, Humphreys MR. Holmium laser enucleation of the prostate (HoLEP): a review and update. Can J Urol. 2019 Aug;26(4 Suppl 1):13-19. PMID 31481144